CLINICAL TRIAL: NCT06032039
Title: Corticosteroid vs Platelet-Rich Plasma Intra-articular Injections in the Treatment of Knee Osteoarthritis in Patients Fifty Years and Older: a Look at Pain and Functional Outcomes at a Single Institution.
Brief Title: Corticosteroid vs Platelet-Rich Plasma Intra-articular Injections in the Treatment of Knee Osteoarthritis.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CREC-MN.023, 2022/2023
Record Dates: First submitted 2023-07-19; First posted 2023-09-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Corticosteroid; Platelet Rich Plasma
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Triamcinolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid Injection (Active Comparator): This arm will receive a corticosteroid (Triamcinalone) injection.
  Interventions: Drug: Triamcinolone
- Platelet Rich Plasma Injection (PRP) (Active Comparator): This arm will receive a PRP injection.
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Drug: Triamcinolone — Standard treatment for osteoarthritis knee pain
  Other Names: Corticosteroid
  Arms: Corticosteroid Injection
Other: Platelet Rich Plasma — Alternative treatment for osteoarthritis knee pain
  Other Names: PRP
  Arms: Platelet Rich Plasma Injection (PRP)

SUMMARY:
This study will explore the effectiveness of intra-articular knee injections in patients with osteoarthritis by comparing Corticosteroid (triamcinolone) vs Platelet Rich Plasma (PRP).

This study is a randomized controlled trial with a sample size of one hundred and sixty patients (160). Patients would be recruited via new referrals and follow-up appointments in the Orthopaedic clinic at the UHWI (University Hospital of the West Indies) with knee osteoarthritis.

The aim of the study is to:

1. To determine if platelet-rich plasma injections are better at improving functional outcomes in the knee using Western Ontario and McMaster Universities Arthritis Index (WOMAC) when compared to intraarticular steroids.
2. To identify adverse reactions related to these injections

DETAILED DESCRIPTION:
This study will explore the effectiveness of intra-articular knee injections in patients with osteoarthritis by comparing Corticosteroid (triamcinolone) vs Platelet Rich Plasma (PRP).

This study is a randomized controlled trial with a sample size of one hundred and sixty patients (160). Patients would be recruited via new referrals and follow-up appointments in the Orthopaedic clinic at the UHWI (University Hospital of the West Indies) with knee osteoarthritis.

The recruitment period will run from July 31, 2023 to January 31, 2024 and a subsequent year of follow-up for each patient.

Selected patients will be informed of the study and given informed consent to fill out once they meet the inclusion criteria. Information will be stored on a password-encrypted external storage device that can only be accessed by the investigator or supervisor. Data will be analyzed using Statistical Package for the Social Sciences (SPSS).

The study will be conducted according to the good clinical practice guidelines of the World Medical Association (WMA) declaration of Helsinki which addresses research on human subjects and will conform to local laws and ethical requirements of the Ministry of Health.

The study will provide information on the effectiveness of two non-operative management of osteoarthritis of the knee; in the form of Platelet-rich plasma and corticosteroid injection. Results from the study can be used as a reference point for future treatment in patients with knee osteoarthritis.

Hypothesis:

PRP is superior to corticosteroid intra-articular injection over one year for knee pain and functional outcome in patients with osteoarthritis of the knee

Design This study is a randomized controlled double-blinded trial. Patients with knee osteoarthritis would be recruited via new referrals and follow-up appointments in the Orthopaedic clinic at the UHWI (University Hospital of the West Indies).

The intervention will be done in the minor operating room at no additional cost to the patient. All the equipment needed will be provided via funding.

* Using the WOMAC scores and visual analogue scale, pain and functional outcomes before and after the procedures will be studied to assess if PRP injection is superior to steroid injection.
* Selected patients will be informed of the study and given an informed consent to fill out once they meet inclusion criteria. Persons consenting will be Orthopaedic residents knowledgeable of the study but will not be a part of the care.
* One person who is not a part of analyzing the data will be in charge of assigning the unique identifying number to each tested knee prior to the start of the study.
* WOMAC questionnaire will be administered at the outpatient clinic visits prior to injection, at two weeks, three months, six months, and a year post-injection.
* Information will be stored on a password-encrypted external storage device that can only be accessed by the investigator or supervisor. Data will be analyzed using Statistical Package for the Social Sciences (SPSS)

Research-related justification for sample size:

The sample size was calculated to be one hundred and sixty patients (160). Calculations for the sample size were done using the formula to calculate the sample size for a two-sample test of means; independent samples T-test. Where:

The type I error rate (5%) The type II error rate (20%)

= The effect size (set at 0.5 for a medium effect size).

Yields a sample size of 64 participants for each group. It is recommended to account for a loss to follow-up of at least 20%, bringing the sample size required for each group to 80, for a total sample size of 160.

Additionally, when considering sample size estimates a larger sample size is always considered better. To estimate a linear regression model to control for other factors such as age and sex, Green (1991) recommends that the sample size should be at least 50 +8*(number of predictors). When seeking to test individual predictors, Green's rule of thumb for a medium effect size is that the sample size be at least 104 + predictors.

Using the estimate of 160, the study should be adequately powered for analysis testing the hypothesis of WOMAC pain scores being different in the group receiving PRP injections compared to the group receiving corticosteroid injection, while controlling for 2 - 3 other characteristics.

Patients will be randomized with the help of an online randomization tool (National Cancer Institute Clinical Trial randomization tool) being placed in one of two arms, corticosteroid vs PRP injection.

Patients will be recruited by the investigator and recruited for the study over 6 months with a further follow-up of up to one year post-injection. The persons assessing the patients at each visit plus the physiotherapist will not be aware of the intervention given.

Patients will be given a single injection of either PRP or corticosteroids (triamcinolone).

All injections will be given by persons post part 1 in the Doctorate of Medicine Orthopaedic program or higher except for the investigators. All patients will have 30 ml of blood taken in an area separate from the location of the centrifuge machine to prepare the PRP.

Patients and administrators will be blinded to the injection by wrapping each syringe before injection. All patients will be injected 20 minutes after the blood has been drawn. The tubes will be sorted by an individual who will know about the desired randomization. Patients will be blinded to the injection as the syringe will be wrapped to hide its content, this will also blind the person administering the injection; who is separate from the person preparing.

The steroid injections are commercially packaged as 40mg/ml. 80 mg of triamcinolone will be used for patients receiving steroids. Preparation of the PRP will be done by the PRP method.

PRP method:

1. Obtain 30mls Whole Blood by venepuncture in acid citrate dextrose (ACD) tubes
2. Do not chill the blood at any time before or during platelet separation.
3. Centrifuge the blood using a 'soft' spin.
4. Transfer the supernatant plasma containing platelets into another sterile tube (without anticoagulant).
5. Centrifuge tube at a higher speed (a hard spin ) to obtain a platelet concentrate.
6. The lower 1/3rd is PRP and upper 2/3rd is platelet- poor plasma (PPP). At the bottom of the tube, platelet pellets are formed.
7. Remove PPP and suspend the platelet pellets in a minimum quantity of plasma (2-4 mL) by gently shaking the tube.

The procedure will be done in the minor operating theatre. Patients will be adequately cleaned with betadine or hibitane in alcohol before venepuncture. Blood will then be brought to a separate sterile room for preparation. Injections will be given under aseptic conditions. The area will be cleaned thoroughly with Povidone-Iodine or Hibitane in 70% Alcohol, depending on the allergy profiles of the patients. With the knee flexed to ninety degrees injection will be given with a 22 gauge needle through the lateral parapatellar space. Dressings will then be applied and patients will be observed for five minutes after the injections, post-procedural analgesics will be given for two days.

Patients will be assessed before injection, at 2 weeks, 3 months, 6 months, and a year post-injection using the WOMAC (Western Ontario and McMaster Osteoarthritis index) and Visual Analogue Score (VAS), by a trained physician who will be blinded to the interventions. There will also be a standardized rehab program for osteoarthritis of the knee developed by the physiotherapy department. This program will be administered for a duration of 6 months to all patients by volunteer registered Physiotherapists in the department.

The proposed start time of the study is July 2023 with the recruitment of patients over 6 months, followed by a one-year follow-up for each patient.

ELIGIBILITY:
Inclusion Criteria:

Kellgren and Lawrence grades 2-3 Age 50 years and older

Exclusion Criteria:

1. Patients with secondary OA:
2. History of Fractures around the knee joint i. patella ii. tibia plateau iii. intra articular distal femur
3. Bleeding diathesis
4. History of septic arthritis
5. Patients on oral steroid medications
6. Patients who received intraarticular steroid injection < 6 months before enrollment
7. Sickle Cell Disease
8. Rheumatoid arthritis
9. Patients with a diagnosis of knee OA with little or no pain
10. Patient with a diagnosis of knee OA being successfully managed with oral medications and physiotherapy
11. Knee pain not attributed to a diagnosis of OA
12. All patients who refuse to participate

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain of the Knee | 1 year of follow up visits, post injection. Follow up will be done at 2 weeks, 3 months, 6 months, and 1 year.
  For pain we are primarily using the visual Analogue scale, which is a subjective pain rating numerical scale where the patients rate their pain on a scale of 0-10.
  The Visual Analogue Scale is a scale from 0-10, where 0 = No Pain and 10 = Worst Pain Possible. The scale also uses faces to indicate the level of pain.
Function of the knee | 1 year of follow up visits, post injection. Follow up will be done at 2 weeks, 3 months, 6 months, and 1 year.
  For Function we are primarily using the Western Ontario and McMaster Universities Arthritis index (WOMAC), which is a commonly used tool to assess pain and function in patients with arthritis. This is a self administered questionnaire with 24 items in 3 subscales (1) 5 points evaluate pain (2) 2 points stiffness (3) 17 points function a numerical score is calculated and used for comparison.
  The WOMAC index uses a scale of 0-4 to rate pain, stiffness and difficulty when doing certain activities, where 0 = None and 4 = Extreme.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Palmer, Principal Investigator — Doctor
Locations (1):
- University Hospital of the West Indies, Kingston, Jamaica

REFERENCES:
- [Background] Forogh B, Mianehsaz E, Shoaee S, Ahadi T, Raissi GR, Sajadi S. Effect of single injection of platelet-rich plasma in comparison with corticosteroid on knee osteoarthritis: a double-blind randomized clinical trial. J Sports Med Phys Fitness. 2016 Jul-Aug;56(7-8):901-8. Epub 2015 Jul 14. PMID 26173792
- [Background] Hirsch G, Kitas G, Klocke R. Intra-articular corticosteroid injection in osteoarthritis of the knee and hip: factors predicting pain relief--a systematic review. Semin Arthritis Rheum. 2013 Apr;42(5):451-73. doi: 10.1016/j.semarthrit.2012.08.005. Epub 2013 Jan 29. PMID 23374502
- [Background] Migliorini F, Driessen A, Quack V, Sippel N, Cooper B, Mansy YE, Tingart M, Eschweiler J. Comparison between intra-articular infiltrations of placebo, steroids, hyaluronic and PRP for knee osteoarthritis: a Bayesian network meta-analysis. Arch Orthop Trauma Surg. 2021 Sep;141(9):1473-1490. doi: 10.1007/s00402-020-03551-y. Epub 2020 Jul 28. PMID 32725315
- [Background] Richards MM, Maxwell JS, Weng L, Angelos MG, Golzarian J. Intra-articular treatment of knee osteoarthritis: from anti-inflammatories to products of regenerative medicine. Phys Sportsmed. 2016;44(2):101-8. doi: 10.1080/00913847.2016.1168272. Epub 2016 Apr 4. PMID 26985986
- [Background] Rayegani SM, Raeissadat SA, Taheri MS, Babaee M, Bahrami MH, Eliaspour D, Ghorbani E. Does intra articular platelet rich plasma injection improve function, pain and quality of life in patients with osteoarthritis of the knee? A randomized clinical trial. Orthop Rev (Pavia). 2014 Sep 18;6(3):5405. doi: 10.4081/or.2014.5405. eCollection 2014 Aug 8. PMID 25317308
- [Background] Gormeli G, Gormeli CA, Ataoglu B, Colak C, Aslanturk O, Ertem K. Multiple PRP injections are more effective than single injections and hyaluronic acid in knees with early osteoarthritis: a randomized, double-blind, placebo-controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):958-965. doi: 10.1007/s00167-015-3705-6. Epub 2015 Aug 2. PMID 26233594
- [Background] Liow Y, Wang W, Loh VW. Outpatient management of knee osteoarthritis. Singapore Med J. 2017 Oct;58(10):580-584. doi: 10.11622/smedj.2017097. PMID 29119193
- [Background] Paik J, Duggan ST, Keam SJ. Triamcinolone Acetonide Extended-Release: A Review in Osteoarthritis Pain of the Knee. Drugs. 2019 Mar;79(4):455-462. doi: 10.1007/s40265-019-01083-3. PMID 30847805
- [Background] Filardo G, Previtali D, Napoli F, Candrian C, Zaffagnini S, Grassi A. PRP Injections for the Treatment of Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Trials. Cartilage. 2021 Dec;13(1_suppl):364S-375S. doi: 10.1177/1947603520931170. Epub 2020 Jun 19. PMID 32551947
- [Background] Green SB. How Many Subjects Does It Take To Do A Regression Analysis. Multivariate Behav Res. 1991 Jul 1;26(3):499-510. doi: 10.1207/s15327906mbr2603_7. PMID 26776715
- [Background] Dhurat R, Sukesh M. Principles and Methods of Preparation of Platelet-Rich Plasma: A Review and Author's Perspective. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):189-97. doi: 10.4103/0974-2077.150734. PMID 25722595